CLINICAL TRIAL: NCT07367672
Title: The Power of Belief: Expectation-driven and Placebo Modulation of Empathic Pain
Acronym: PoB-EP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Weihua Zhao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-102
Record Dates: First submitted 2025-12-26; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Analgesic expectation; Empathic pain; fMRI; Oxytocin; Placebo

STUDY DESIGN:
Intervention Model Description: The placebo (PLC) and oxytocin (OXT) spray conditions were conducted under a single-blind design due to all participants in both the placebo and oxytocin conditions will be informed that they are receiving oxytocin, described as a potent agent for pain relief.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The placebo (PLC) and oxytocin (OXT) spray conditions were conducted under a single-blind design due to all participants in both the placebo and oxytocin conditions will be informed that they are receiving oxytocin, described as a potent agent for pain relief.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intranasal Oxytocin (Active Comparator): Administer oxytocin (24 IU) intranasally.
  Interventions: Drug: Intranasal Oxytocin (OT) 24 IU
- Intranasal placebo (Active Comparator): Administer placebo intranasally.
  Interventions: Drug: Intranasal placebo administration
- Intranasal nothing (control) (No Intervention): Control condition

INTERVENTIONS:
Drug: Intranasal Oxytocin (OT) 24 IU — Administer oxytocin (24 IU) intranasally, 6 individual 0.1 ml puffs (4 IU/0. 1ml), three puffs per nostril one every 30 seconds. The participants will be informed that they are receiving oxytocin, described as a potent agent for pain relief.
  Other Names: Intranasal Oxytocin
  Arms: Intranasal Oxytocin
Drug: Intranasal placebo administration — Administer placebo intranasally, 6 individual 0.1 ml puffs, three puffs per nostril one every 30 seconds. The participants will be informed that they are receiving oxytocin, described as a potent agent for pain relief.
  Other Names: Intranasal placebo
  Arms: Intranasal placebo

SUMMARY:
This study investigates how belief and expectation influence empathic pain-the pain we feel when observing others in distress. Healthy adult participants will be randomly assigned to one of three groups: no-treatment control, placebo nasal spray, oxytocin-containing nasal spray. Participants in both the placebo and oxytocin conditions will be informed that they are receiving oxytocin, described as a potent agent for pain relief. During functional MRI scanning, all participants will view naturalistic pain-related videos and provide ratings of perceived subjective pain. The study aims to examine how cognitive beliefs and neuromodulatory interventions alter subjective pain experience and brain activity, including changes in brain network communication.

DETAILED DESCRIPTION:
This study examines how belief-driven expectations modulate empathic pain at both behavioral and neural levels. Healthy adult participants will be randomly assigned to one of three groups: no-treatment control, placebo nasal spray, oxytocin-containing nasal spray. Participants in both the placebo and oxytocin conditions will be informed that they are receiving oxytocin, described as a potent agent for pain relief.

During fMRI scanning, participants will complete a naturalistic empathic pain task by viewing videos depicting others in pain and rating their perceived pain on a standardized scale. Behavioral data will be transformed into analgesia-weighted scores to capture individual sensitivity to expectation-driven analgesia. Neural data will include whole-brain voxel-wise activity, multivariate predictive patterns derived from partial least squares regression (PLSR), and directed functional connectivity assessed using lagged partial-correlation directionality analysis (LPC-DA) to evaluate top-down and bottom-up information flow.

The primary objectives are to (1) assess the behavioral effects of expectation-driven analgesia, (2) identify brain regions predictive of pain modulation, and (3) characterize hierarchical network reorganization under different interventions.

ELIGIBILITY:
Inclusion Criteria:

* (1) Healthy subjects without any past or present psychiatric or neurological disorders; (2) Healthy subjects without any current psychotherapeutic medication.

Exclusion Criteria:

* (1) Participant with any past or present psychiatric or neurological disorders; (2)Participant with any current psychotherapeutic medication.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on biological sex. Both male and female participants are eligible. Female participants must confirm that they are not pregnant, not using hormonal contraceptives, and not menstruating during the study period.
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Analgesia-weighted empathic pain ratings (R') | During fMRI scanning (45 minutes follollowing treament adminstration), for each video stimulus presentation
  Subjective pain ratings for each stimulus adjusted for treatment-specific baseline and analgesia-dependent gain to capture individual sensitivity to expectation-driven analgesia.
Whole-brain multivariate predictive patterns | During fMRI scanning (45 minutes follollowing treament adminstration), analyzed post-session
  Partial least squares regression (PLSR) will be applied to voxel-wise fMRI contrast maps to identify latent components that predict analgesia-weighted pain scores under different interventions.
Directed functional connectivity and network hierarchy | During fMRI scanning (45 minutes follollowing treament adminstration), analyzed post-session
  Lagged partial-correlation directionality analysis (LPC-DA) among key regions identified by PLSR will quantify top-down and bottom-up information flow in empathic pain circuits.

CONTACTS AND LOCATIONS:
Overall Officials: Siying Wang, Study Chair — University of Electronic Science and Technology of China
Locations (2):
- China (2):
  - Weihua Zhao, Chengdu, Sichuan
  - University of Electronic Science and Technology of China, Chengdu

IPD SHARING:
Plan to Share IPD: No